CLINICAL TRIAL: NCT00530322
Title: Adhesion Formation Following Laparoscopic and Open Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Other Study IDs: 06/Q1909/68
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Adhesions
Keywords: Adhesions; Laparoscopy; Colorectal surgery; Colorectal disease
MeSH Terms: conditions — Tissue Adhesions | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients who have had previous open colorectal surgery and are referred for a further operative procedure, at which time a "second-look" laparoscopy can be performed.
  Interventions: Procedure: Laparoscopy
- B: Patients who have had a previous laparoscopic colorectal procedure and are having a "second-look" procedure
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — A "second-look" laparoscopy, in patients who require further surgery (for example a liver resection or closure of ileostomy).

SUMMARY:
To ascertain whether there are fewer adhesions (internal scars) formed following laparoscopic (key-hole) surgery for colorectal diseases than traditional open surgery.

ELIGIBILITY:
Inclusion Criteria:

* Previous elective colonic or rectal resection
* Having a further operative intervention at which time a laparoscopy can be performed

Exclusion Criteria:

* Children <18
* Further surgery not relating to the primary colorectal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-06; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Rockall, FRCS, Study Director — The Royal Surrey County Hospital
Locations (1):
- The Royal Surrey County Hospital, Guildford, Surrey, United Kingdom